CLINICAL TRIAL: NCT06645171
Title: Effect of an Oral Nutritional Supplement (ONS) with Prebiotic Fibre Compared to a Non-fibre Containing ONS Equal in Energy and Protein Content on Gut Microbiota Bifidobacteria in Older Adults with or At Risk of Disease Related Malnutrition
Brief Title: Effect of an Oral Nutritional Supplement (ONS) with Prebiotic Fibre Compared to a Non-fibre Containing ONS Equal in Energy and Protein Content on Gut Microbiota in Older Adults with or At Risk of Disease Related Malnutrition
Acronym: BISON
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 23REX0060367
Record Dates: First submitted 2024-10-10; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Changes in Gut Microbiota Bifidobacterial Levels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): ONS including fibre (300 kcal, 12gr protein, 125 mL, 4.5 g fibre), The subjects will use study products twice daily for 4 weeks starting at V1.
  Interventions: Dietary Supplement: Fibre drink
- Arm 2 (Experimental): ONS without fibre (300 kcal, 12gr protein, 125 mL, 0 g fibre), The subjects will use control products twice daily for 4 weeks starting at V1.
  Interventions: Dietary Supplement: Fibre drink

INTERVENTIONS:
Dietary Supplement: Fibre drink — One drink will be tested

SUMMARY:
This study assesses the effects of an oral nutritional supplement (ONS) with fibre compared to a non-fibre containing ONS equal in energy and protein content on gut microbiota bifidobacteria in older adults with or at risk of disease related malnutrition. It is a randomised controlled, double blind, parallel-group, multi-country study. Subjects will receive an ONS with or without (control group) fibre. They take it twice a day for 4 weeks and the change in their gut microbiota bifidobacterial levels is the primary outcome. They will be measured at day 1 (V1), day 15 (V2) and week 4 (V3).

ELIGIBILITY:
Inclusion Criteria:

* 1. 65 years of age or older 2. Identified as at medium or high risk of malnutrition based on:

  a) MNA-SF score between 0 - 11 and / or b) are prescribed with ONS 3. In need of 2 servings of oral nutritional support/day (300 kcal; 12 gr protein per serving).

  4. a) Not being prescribed with ONS or b) being prescribed with non-fibre containing ONS and willing and able to switch from pre-study prescribed ONS to the Test or Control Product for participation in the study.

  5. Willing to maintain dietary habits for the duration of the study. Written informed consent from subject (or impartial witness after verbal consent of subject when subject is physically unable to sign and where allowed by local regulations).

Exclusion Criteria:

* 1. Requirement for a fibre-free diet. 2. Have used nutritional supplements with fibre/prebiotics and/or probiotics content at any point during 3 weeks prior to start study (Visit 1) and / or will not refrain from using these kinds of products during the study period.

  3. Admitted to an intensive care unit. 4. Hemodynamically unstable. 5. Known allergy to cow's milk protein. 6. Known galactosaemia. 7. Known hepatic encephalopathy. 8. Known Irritable Bowel Syndrome. 9. Known severe lactose intolerance without using lactase. 10. Known history of GI surgery. 11. Known history of intestinal polyp removal within 3 months prior to the study.

  12. Known history of Immunotherapy. 13. Known history of GI cancer. 14. Active cancer treatment or within 12 months prior the study 15. Diagnose of Celiac Disease. 16. Received antibiotics within 4 weeks prior to study. 17. Patients following a vegan or vegetarian diet. 18. Active flare of inflammatory bowel disease as defined by HBI >6 (Crohn's disease) or SCCAI >5 (ulcerative colitis).

  19. Stricturing Crohn's disease. 20. Any contraindication to oral feeding per se being: gastrointestinal failure or suppressed gastrointestinal function, complete intestinal obstruction and major intra-abdominal sepsis.

  21. Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements, for example due to the presence of a psychiatric disorder (e.g. major depression, psychoses), dementia or Alzheimer's disease.

  22. Planned hospital admission during the study period in case not hospitalised at screening 23. Participation in any other studies involving investigational or marketed products concomitantly or within 6 weeks prior to baseline.

  24. Severe disease with life expectancy less than a year.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in gut microbiota bifidobacterial levels | 4 weeks

SECONDARY OUTCOMES:
Changes in gut microbiota composition | 4 weeks
Fecal pH | 4 weeks
Stool frequency and consistency assessed by the Bristol Stool Form Scale (BSFS) | 4 weeks
Total short-chain fatty acids (SCFA) | 4 weeks